CLINICAL TRIAL: NCT01235104
Title: Impact of Total Nephrectomy on Patients With Kidney Stone
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Alexandre Danilovic, Urology Department
Other Study IDs: 0652/10
Record Dates: First submitted 2010-11-03; First posted 2010-11-05 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2001-01

CONDITIONS: Kidney; Urolithiasis; Nephrectomy; Treatment Outcome; Complications
MeSH Terms: conditions — Urolithiasis | interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total nephrectomy
  Interventions: Procedure: Total nephrectomy

INTERVENTIONS:
Procedure: Total nephrectomy — Total nephrectomy

SUMMARY:
The aim of this study is to investigate the outcomes of total nephrectomy on patients with kidney stone disease.

DETAILED DESCRIPTION:
The aim of this study is to retrospectively investigate the effects of total nephrectomy on renal function, quality of life, early and late complications and development of the stone disease on the remnant unit on patients with kidney stone disease.

ELIGIBILITY:
Inclusion Criteria:

* Total nephrectomy
* Kidney stone disease

Exclusion Criteria:

* < 18 y.o.
* Cancer
* Kidney transplant
* Solitary kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with kidney stone submitted to total nephrectomy from january 2001 to october 2010 at University of Sao Paulo General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2001-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Danilovic, M.D., Ph. D., Principal Investigator — Department of Urology of University of Sao Paulo General Hospital